CLINICAL TRIAL: NCT01302600
Title: Phase II, Multicenter, Randomized, Adaptive, Double-blind, Placebo Controlled Study to Assess Safety and Efficacy of Olesoxime (TRO19622) in 3-25 Year Old Spinal Muscular Atrophy (SMA) Patients.
Brief Title: Safety and Efficacy of Olesoxime (TRO19622) in 3-25 Years SMA Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Association Française contre les Myopathies (AFM), Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WN29836; TRO19622 CL E Q 1275-1 (Other: Trophos ID)
Record Dates: First submitted 2011-02-18; First posted 2011-02-24 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Spinal Muscular Atrophy Type II; Spinal Muscular Atrophy Type III Non Ambulant
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood | interventions — olesoxime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olesoxime (Experimental): 100 patients in this arm. liquid suspension
  Interventions: Drug: Olesoxime
- Placebo (Placebo Comparator): 50 patients enrolled in this arm. liquid suspension
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olesoxime — Liquid suspension formulation, 100 mg/ml at a dose of 10 mg/kg will be administered once a day with food at dinner
  Arms: Olesoxime
Drug: Placebo — 0.1ml/kg once a day with food at dinner.
  Arms: Placebo

SUMMARY:
Assess the efficacy and the safety of olesoxime in SMA type 2 or type 3 non ambulant patients aged 3-25 years

DETAILED DESCRIPTION:
This study is a multicenter, double-blind, randomized, adaptive, parallel groups, placebo controlled 3-stage study in patients with SMA type 2 or non ambulant type 3.

Stage 1 DMC 3-month safety assessment: An independent Data Monitoring Committee (DMC)will assess the safety of olesoxime every 3 months.

Stage 2 Efficacy/futility analyses at one year: A first interim efficacy analysis will be performed after all patients have been treated for one year (52 weeks) in order to assess the need to continue the study to reach the planned objective. In the event of positive and significant results in favor of olesoxime, the study will be considered as successful and all patients will be switched to olesoxime to allow the assessment of the sustainability of the treatment effect and safety. If the results are significantly in favor of placebo, the study will be discontinued for failure (futility).

Stage 3 Efficacy and safety analysis at two years: The expected study duration is of 2 years (104 weeks) to show efficacy. If the study is not discontinued for futility or medication regimen is changed due to success, the study will therefore continue until planned completion i.e. 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Weakness and hypotonia consistent with a clinical diagnosis of spinal muscular atrophy (SMA) type II or III
* Laboratory documentation of homozygous absence of SMNI exon 7 and/or deletion and mutation on other allele
* MFM relative score (percentage of the maximum sum of both dimensions) >= 15% (D1 + D2 score)
* HFMS score at baseline >= 3
* Non ambulant patients defined as patients with HFMS score =< 38
* Must be 3 years of age or older, but younger than 26 years of age, at time of enrolment
* Age of onset of symptoms =< 3 years of age
* Signed informed consent of patient and/or parents/guardian
* Laboratory results drawn within 31 days prior to start of study entry demonstrating no clinically significant abnormalities
* Ability to take the study treatment (tested at screening after informed consent)

Exclusion Criteria:

* Evidence of renal dysfunction, blood dysplasia, hepatic insufficiency, symptomatic pancreatitis, congenital heart defect, known history of metabolic acidosis, hypertension,significant central nervous system impairment, or neurodegenerative or neuromuscular disease other than SMA
* Any clinically significant ECG abnormality
* Any acute co-morbid condition interfering with the well-being of the subject within 7 days of enrolment including bacterial infection, viral infectious processes, food poisoning, temperature > 37.0 °C, the need for acute treatment or observation due to any other reason, as judged by the investigator; patient can be included after resolution of the acute event
* Use of medications intended for the treatment of SMA including riluzole, valproic acid, hydroxyurea, sodium phenylbutyrate, butyrate derivatives, creatine, carnitine, growth hormone, anabolic steroids, probenecid, oral or parenteral use of corticosteroids at entry, agents anticipated to increase or decrease muscle strength or agents with known or presumed histone deacetylase (HDAC) inhibition, within 30 days prior to study entry. Subjects who use a nebulizer or require an inhaler to steroids will be allowed in the study; however oral use of steroids is prohibited. The oral use of salbutamol is permitted with the following restrictions: patients should have been on salbutamol for at least 6 months before inclusion in the trial, with good tolerance. The dose of salbutamol should remain constant for the duration of the trial. The use of inhaled beta-agonists (for the treatment of asthma crisis for example) is allowed.
* Spinal rod or fixation for scoliosis within the past 6 months or anticipated need of rod or fixation within 6 months of enrolment.
* Inability to meet study visit requirements or cooperate reliably with functional testing
* Coexisting medical conditions that contraindicate travel, testing or study medications
* Olesoxime is contraindicated in subjects/patients who develop drug hypersensitivity to it or one of the formulation excipients including hypersensitivity to sesame oil.
* Patients with hemostasis disorders
* Patients with known biliary tract obstruction
* Current or planned pregnancy or nursing period
* For Women: Failure to use one of the following safe methods of contraception:

  1. Female condoms, diaphragm or coil, each used in combination with spermicides
  2. Intra-uterine device
  3. Hormonal contraception in combination with a mechanical method of contraception
* Participation in any other investigational drug or therapy study within the previous 3 months.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 165 (Actual)
Dates: Start 2010-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Motor Function Measure | every 6 months
  Motor function Measure (MFM) D1+D2 score

SECONDARY OUTCOMES:
responder analyses on MFM and HFMS, time to 4 point decrease on HFMS, CMAP/MUNE, PedsQL, FVC, CGI and safety | every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Bertini, MD, Principal Investigator — Bambino Gesu Hospital
Locations (22):
- Belgium (2):
  - University Hospitals, Ghent
  - University Hospitals, Leuven
- France (6):
  - Hôpital Femme-Mère-Enfant, Bron
  - Hôpital Raymond Poincaré, Garches
  - CHRU Hôpital R. Salengro, Lille
  - Hôpital La Timone, Marseille
  - CHU de Montpellier, Hôpital Gui de Chauliac, Montpellier
  - Groupe hospitalier Armand-Trousseau, Paris
- Germany (3):
  - University of Essen, Essen
  - Universitat Klinikum Freiburg, Freiburg im Breisgau
  - Friedrich-Baur-Institute, München
- Italy (6):
  - Istituto Giannina Gaslini, Genova
  - AOU Policlinico, Messina
  - Centro Dino Ferrari, Milano, Milan
  - NEuroMuscular Omnicentre (NEMO), Milan
  - Bambino Gesu' Research Children's Hospital, Roma
  - Policlinico Universitario "Agostino Gemelli",, Roma
- University Medical Center, Utrecht, Netherlands
- Medical University of Warsaw, Warsaw, Poland
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Birmingham
  - Dubowitz Neuromuscular Centre, London
  - Institute of Human Genetics, Newcastle

REFERENCES:
- [Derived] Bertini E, Dessaud E, Mercuri E, Muntoni F, Kirschner J, Reid C, Lusakowska A, Comi GP, Cuisset JM, Abitbol JL, Scherrer B, Ducray PS, Buchbjerg J, Vianna E, van der Pol WL, Vuillerot C, Blaettler T, Fontoura P; Olesoxime SMA Phase 2 Study Investigators. Safety and efficacy of olesoxime in patients with type 2 or non-ambulatory type 3 spinal muscular atrophy: a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Neurol. 2017 Jul;16(7):513-522. doi: 10.1016/S1474-4422(17)30085-6. Epub 2017 Apr 28. PMID 28460889